CLINICAL TRIAL: NCT00368329
Title: Phase I Study of Dose Escalation Using Image-guided Radiotherapy to Deliver a Stereotactic Radiosurgical Boost After Neoadjuvant Chemoradiotherapy in Patients With Locally Advanced Esophageal Cancer
Brief Title: Phase I Dose Escalation of Stereotactic Radiosurgical Boost for Locally Advanced Esophageal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel T. Chang, PI, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESOPH0001; 96075 (Other: Stanford University Alternate IRB Number)
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma | interventions — Capecitabine; Fluorodeoxyglucose F18; Fluorouracil; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — PO bid daily on RT days: 500mg & 150mg tabs for dose 825mg/m2 bid AM/PM (total daily dose 1650mg/m2)
  Other Names: Xeloda
Drug: [18-F] Fluorodeoxyglucose (FDG) — 5-10 mCi IV administration
  Other Names: Fluorodeoxyglucose
Drug: 5-Fluorouracil (5-FU) — 200mg/m2 continuous venous infusion
  Other Names: 5-Fluorouracil; Carac; Efudix; Efudex; Fluoroplex
Drug: Carboplatin — AUC 2, based onCalvert formula IV infusion
  Other Names: cis-Diammine; Paraplatin; Paraplatin-AQ

SUMMARY:
To study the safety and feasibility of stereotactic radiation dose escalation following neoadjuvant chemotherapy with concurrent conventionally fractionated radiation, by evaluating the acute and late toxicity of treatment.

DETAILED DESCRIPTION:
This study will evaluate the safety and feasibility of delivering radiation dose escalation using hypofractionated radiosurgery in locally advanced esophageal cancer. The dose escalation will be delivered using an image-guided radiosurgical boost to the tumor volume, following a neoadjuvant regimen consisting of oxaliplatin, capecitabine, and conventionally fractionated radiotherapy. In addition, we will evaluate the utility of PET-FDG before and after neoadjuvant chemoradiation in predicting the pathologic response to pre-operative treatment. We will study the effect of this regimen on pathologic complete response rates and complete resection rates at surgery among patients with locally advanced esophageal cancer and determine patterns of failure and rates of progression-free survival. Finally, we plan to characterize in an exploratory manner the correlation between molecular markers and pathologic findings following pre-operative chemoradiation.

ELIGIBILITY:
Inclusion Criteria:- Confirmed diagnosis of adenocarcinoma or squamous cell carcinoma of the esophagus by pathologist.

* Endoscopic ultrasound or CT evidence of tumor penetration through the esophageal wall or involvement of regional lymph nodes, without evidence of distant metastasis
* No prior chest radiation therapy
* No prior chemotherapy for esophageal cancer
* Age greater than 18 years
* No infections requiring antibiotic treatment
* Able to care for self
* Patients must have acceptable liver, kidney and bone marrow function.
* The effects of the chemotherapy drugs on the developing human fetus are unknown. Women of child-bearing potential and men must agree to use adequate contraception. Exclusion Criteria:- Patients receiving any other investigational agents
* Evidence of distant metastases
* Uncontrolled medical illness
* Any malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix.
* Pregnant and breastfeeding women are excluded.
* HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
A complete assessment of all pathologic specimens (biopsy and definitive surgical) to document the histology, grade, depth of invasion, lymphovascular or perineural invasion.
The inked margins on the definitive surgical specimen will be inked and margin status, size of the tumor, evidence of residual tumor will be recorded.
Patients' responses to therapy will be evaluated clinically after completion of their neoadjuvant chemoradiation. | after completion of their neoadjuvant chemoradiation

SECONDARY OUTCOMES:
Physical exam | Once every three months for two years, then every six months for three years and then once a year.
CT scan | Three months after completion of therapy, then every six months for three years then once a year for until 5 years from completion of therapy.
Upper endoscopy | Three months after completion of therapy, then every six months for three years then once a year for until 5 years from completion of therapy.
Patterns of failure and the 2-year progression-free survival (PFS) rate. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Chang, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States